CLINICAL TRIAL: NCT01616771
Title: GlideScope®Video Laryngoscope for Difficult Intubation: Implication of the Size of Blade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: H-1111-037-385
Record Dates: First submitted 2012-04-30; First posted 2012-06-12 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Intubation; Difficult
Keywords: laryngoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- glottis view assessment (Other): Glottis view assessment using Macintosh laryngoscope & GVL selected by weight & smaller sized GVL in single patient
  Interventions: Device: Macintosh laryngoscope; Device: GVL selected by weight; Device: smaller sized GVL

INTERVENTIONS:
Device: Macintosh laryngoscope — Glottis view assessment by direct visualization using Macintosh laryngoscope
Device: GVL selected by weight — Glottis view assessment by GVL selected by weight which is usually selected first
  Other Names: GlideScope® videolaryngoscopy selected by weight
Device: smaller sized GVL — Glottis view assessment by GVL which is smaller in one size than GVL selected by age
  Other Names: smaller sized GlideScope® videolaryngoscopy

SUMMARY:
The investigators evaluated the usefulness of the Glidescope(GVL) compared with direct laryngoscopy in patients whose airway management are anticipated difficult (C&L grade ≥3) by comparing the laryngoscopic view. Also, the investigators compared the effectiveness of smaller-size blade of GVL (GVLs) with standard blade of GVL selected by patient's weight (GVLw) in the same patients.

DETAILED DESCRIPTION:
We assumed that smaller sized GVL can slide more angulated along the tongue, so the tip of a blade can be placed more anterior and cephalad. The angle of camera would be optimized by inserting the blade further with the blade tip directed toward the larynx. This optimization may be more remarkable with smaller blade because it can be inserted with rotation. Furthermore, the location and the angle of camera are different according to GVL blade size. Considering that patient with difficult airway has hypognathia and more cephalad larynx, it may be helpful with smaller sized GVL (GVLs) rather than GVL selected by weight (GVLw) for improvement of laryngoscopic view in patients with difficult airways. We hypothesized that GVLs can provide better laryngoscopic view than GVLw and DL in patient with difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose C&L grade were over 3 in previous anesthetic records.

Exclusion Criteria:

* Patients with pulmonary aspiration, increased intracranial pressure, and severe cardiovascular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, professor, Study Director — Seoul National University Hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- Glottis View Assessment: After checking the C&L grade using Macintosh laryngoscope, C&L grade was re-evaluated using GVL selected by weight and smaller sized GVL in consecutive order.
Period: Macintosh Laryngoscopy for 5 Sec
Arm/Group | Glottis View Assessment
Started | 23
Completed | 23
Not Completed | 0
Period: GVL Selected by Weight for 5 Sec
Arm/Group | Glottis View Assessment
Started | 23
Completed | 23
Not Completed | 0
Period: Smaller Sized GVL for 5 Sec
Arm/Group | Glottis View Assessment
Started | 23 (Four of 23 patients could not be evaluated by smaller sized GVL, because there was no smaller one.)
Completed | 19
Not Completed | 4
Not completed — lack of GVL size | 4

BASELINE CHARACTERISTICS:
Arm/Group | Glottis View Assessment
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: The Differences in the Glottis View (C&L Grade) of Macintosh Laryngoscope and GVL Selected by Weight.
Description: Glottis view was scored using C&L grade by Macintosh laryngoscope and GVL selected by weight, and compared each other.
  We used modified C&L grade: grade 1, all or most of the glottic aperture was visible; grade 2a, posterior cords and cartilage visible; grade 2b, only posterior cartilage visible; grade 3a, epiglottis visible and can be lifted; grade 3b, epiglottis adherent to the posterior pharynx; and grade 4, the epiglottis could not be visualized.
  For the statistical analysis, the modified C&L grade was converted to an ordinal scale; grade 1 to 1, grade 2a to 2, grade 2b to 3, grade 3a to 4, grade 3b to 5, and grade 4 to 6. Therefore, score range for the data reported in the table was between 1 and 6, with 1 representing best view and 6 representing no view.
Time Frame: up to 1 day of surgery
Measure: Median (95% Confidence Interval); unit: units on a scale
Groups:
- Macintosh Laryngoscope: After induction of anesthesia, Macintosh laryngoscope was inserted into mouth and C&L grade was checked.
- GVL Selected by Weight: Right after Macintosh laryngoscope was removed, C&L grade was reassessed by second laryngoscopy, using GVL selected by weight.
Arm/Group | Macintosh Laryngoscope | GVL Selected by Weight
Number analyzed (Participants) | 23 | 23
units on a scale | 6 [5.5 to 6] | 5.5 [5 to 6]
Statistical Analysis 1: Comparison: Macintosh Laryngoscope vs GVL Selected by Weight; An improvement of C&L grade ordinal scale by 2 was considered a clinically significant change. The mean difference of C&L grade ordinal scale between DL and GVLw was 1.3, and its standard deviation was 2.0 in our pilot study. The required sample size for the Wilcoxon signed rank test was 21 with an α error of 0.05 and 80% power; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — To verify the difference in C&L grades using each blade, the ordinal scales of each blade were compared using the Wilcoxon signed rank test. P values and confidence intervals have been corrected for the 3 comparisons; Hodges-Lehmann method was used to calculate 98.3% CIs of paired differences of 3 comparisons

2. Secondary Outcome: The Differences in the Glottis View (C&L Grade) of GVL Selected by Weight and Smaller Sized GVL
Description: Glottis view was scored using C&L grade by GVL selected by weight and smaller sized GVL, and compared each other.
  Score range for the data reported in the table was between 1 and 6, with 1 representing best view and 6 representing no view.
Time Frame: up to 1day of surgery
Population: Four of 23 patients could not be evaluated by smaller sized GVL because there was no smaller blade than their GVL selected by weight.
Measure: Median (95% Confidence Interval); unit: units on a scale
Groups:
- Smaller Sized GVL: The C&L grade was reassessed by smaller sized GVL, after removal of GVL selected by weight
Arm/Group | GVL Selected by Weight | Smaller Sized GVL
Number analyzed (Participants) | 23 | 19
units on a scale | 5.5 [5 to 6] | 1 [1 to 1.5]
Statistical Analysis 1: Comparison: GVL Selected by Weight vs Smaller Sized GVL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; Hodges-Lehmann method was used to calculate 98.3% CIs of paired differences of 3 comparisons

ADVERSE EVENTS:
Time Frame: up go 1 days after surgery
Groups:
- Macintosh Laryngoscope: C&L grade assessment by Macintosh laryngoscope, after induction of anesthesia
- GVL Selected by Weight: C&L grade assessment by GVL selected by weight, after removal of Macintosh laryngoscope
- Smaller Sized GVL: C&L grade assessment by smaller sized GVL, after removal of GVL selected by weight
Arm/Group | Macintosh Laryngoscope | GVL Selected by Weight | Smaller Sized GVL
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No